CLINICAL TRIAL: NCT01550978
Title: The Safety of Using the AnapnoGuard 100 System in Intubated Critical Care Patients
Brief Title: Evaluation of the Safety and Efficacy of the AnapnoGuard 100 System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitech Respiration (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HST-AG-04
Record Dates: First submitted 2012-02-21; First posted 2012-03-12 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Intubation Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): Patients intubated with AnapnoGuard EndoTracheal Tube and connected to the AnapnoGuard 100 Control System
  Interventions: Device: AnapnoGuard 100 System
- Control Group (No Intervention): Patients intubated with the Standard of Care EndoTracheal Tube and Connected to a Suction Regulator

INTERVENTIONS:
Device: AnapnoGuard 100 System — AnapnoGuard™ 100 Respiratory Guard System is intended for airway management by oral/nasal intubation while providing continuous endotracheal cuff pressure control using non-invasive measurement and monitoring of carbon dioxide concentration in the subglottic space and evacuation of secretions from above the endotracheal tube's cuff.
  Arms: Study Group

SUMMARY:
The purpose of this study is to evaluate the safety of using the AnapnoGuard 100 system during the course of mechanical ventilation and intubation of critical care patients in Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Age above 21 (men and women);
* Patient is admitted to ICU and expected to receive mechanical ventilation for more than 12 hours
* Absence of clear signs of pneumonia and lung contusion on chest X ray;
* For study patients, connection of the ETT to the AnapnoGuard system less than 6 hours from intubation initiation;
* No fever or fever from a known non chest/lung origin;

Exclusion Criteria:

* Patients who had been treated with mechanical ventilation during the last 3 months;
* Patients with facial, oropharyngeal or neck trauma
* BMI > 40
* Pregnant women
* Patients ventilated in prone position
* Difficult intubation (defined as more than 3 intubation attempts)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Rate of AE (adverse events) and SAE (serious adverse events) | participants will be followed for the entire duration of intubation (an expected average of 8 days)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, Prof., Principal Investigator — Director of General ICU and Institute of Anesthesiology and Intensive Care, Policlinico Universitario A. Gemelli
Locations (1):
- Policlinico Universitario A. Gemelli, Rome, Italy

REFERENCES:
- [Derived] De Pascale G, Pennisi MA, Vallecoccia MS, Bello G, Maviglia R, Montini L, Di Gravio V, Cutuli SL, Conti G, Antonelli M. CO2 driven endotracheal tube cuff control in critically ill patients: A randomized controlled study. PLoS One. 2017 May 11;12(5):e0175476. doi: 10.1371/journal.pone.0175476. eCollection 2017. PMID 28493877